CLINICAL TRIAL: NCT05316987
Title: Effect of Narrow Band Ultraviolet B on the Tissue Level of Interleukin 15 and Interleukin 15 Receptor Alpha Subunit in Active Non Segmental Vitiligo Cases.
Brief Title: Effect of NB-UVB on the Tissue Level of IL 15 and IL-15Rα in Active Non Segmental Vitiligo Cases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Emad, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS_ 270_2021
Record Dates: First submitted 2022-02-18; First posted 2022-04-07 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Active Non Segmental Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active vitiligo patients (Other): NBUVB
  Interventions: Radiation: Narrow band ultraviolet B

INTERVENTIONS:
Radiation: Narrow band ultraviolet B — 48 sessions of narrow band ultraviolet

SUMMARY:
This study aims at evaluating the effect of NB-UVB on tissue level of IL-15 and IL-15 receptor alpha subunit (IL-15Rα)(CD215) in active non segmental vitiligo. This in turn will shed light on the potential role of phototherapy as a safe mean of prevention of vitiligo recurrence as well as evaluating the utility of IL 15 and IL 15 Rα as markers of vitiligo activity/recurrence.

DETAILED DESCRIPTION:
Vitiligo is a T cell-mediated, autoimmune cutaneous disorder characterized by loss of functioning melanocytes from the basal layer of epidermis and/or hair follicles, leading to depigmented areas of the skin, mucous membranes, and/or hair (Strassner et al., 2018).

Multiple factors have been involved in disease development, with a prominent role of the immune system, in particular T cells. After repigmentation, vitiligo usually recurs in the same area, drawing attention to the fact that resident memory T cells (TRM) are present at the sites of vitiligo lesions. This was confirmed by a number of studies (Boniface et al., 2018 , Boniface& Seneschal., 2019 , Riding& Harris., 2019) showing that stable and active vitiligo perilesional skin is enriched with a population of CD8 TRM expressing both CD69 and CD103. CD8 TRM expressing CD103 are localized mainly in the epidermis. IL-15 is the only identified cytokine required for maintenance of CD8 TRM cells (Baumann et al., 2018 and Richmond et al., 2018).

Interleukin 15(IL-15) is one of Interleukin 2(IL-2) family members. It plays an important function in the pathogenesis of multiple cutaneous autoimmune diseases as psoriasis (Rückert et al.,2000) , alopecia areata (Ebrahim et al.,2019) and vitiligo (Atwa et al.,2020).

IL-15 receptor (IL-15R) is expressed on natural killer cells, dendritic cells, monocytes, fibroblasts, T cells and keratinocytes . IL-15R is composed of α (CD215), β (CD122), and γ (CD132) chains , The alpha chain occurs as both a soluble and a membrane-attached subunit (Vámosi et al., 2004 , Budagian et al., 2006 and Di Sabatino et al.,2011).

IL-15 stimulates neighbor cells by a trans-presentation mechanism through secretion of (IL-15. IL-15Rα complexes) from the surface of monocytes or dendritic cells into endosomes for its presentation in trans to neighboring cytotoxic cells or Natural killer cells ( Stonier & Schluns .,2010).

IL-15 enhances maturation and survival of natural killer (NK) cells, neutrophils, and Dendritic cells (DCS) (Di Sabatino et al.,2011). Additionally, IL-15 promotes NK cell cytotoxicity and cytokine production such as interferon gamma( IFN-γ )and tumour necrosis factor alfa (TNF-α) (Fehniger & Caligiuri .,2001). As for DCs, they regulate the development and survival of memory cytotoxic cells by IL-15 trans-presentation ( Budagian et al., 2006 and Stonier & Schluns.,2010). Furthermore, IL-15 promotes T-cell receptor-dependent proliferation of Th17 (Di Sabatino et al.,2011).

TRM primarily express the CD122 (IL-15R β) subunit, a shared component of the receptors for IL-2 and IL-15, whereas keratinocytes express more CD215(IL-15Rα) in lesional compared to non lesional skin which is consistent with an ability to present IL-15 to T cells in trans (Richmond et al., 2018).

CD122(IL-15R β) expression is significantly higher on melanocyte-specific T cells in both mouse and human vitiligo compared to endogenous memory T cells, suggesting that autoreactive T cells are more dependent on IL-15 than non-autoreactive T cells. In addition, anti-CD122 blocking antibody inhibit IL-15 mediated T cell survival but not IL-2-mediated proliferation in vitro. This is consistent with the role of IL-15 in mediating T cell survival, but not proliferation (Riding et al., 2018).

These findings are consistent with an important role of IL-15 in maintenance of autoreactive TRM cells in vitiligo and suggest that this could be an effective targeted treatment strategy for vitiligo patients ( Frisoli et al., 2020).

Phototherapy has been considered as a cornerstone in management of vitiligo patients (Esmat et al., 2017). Narrow band ultraviolet B (NB-UVB) has been found to be an effective and well-tolerated treatment option in vitiligo compared to other available photo(chemo)therapy options (Sokolova et al., 2015).

Regarding effect of Ultraviolet B treatment on IL-15 in normal skin, it was found to increase IL-15 expression in epidermal and dermal sheets as well as in cultured keratinocytes and dermal fibro-blasts (Mohamadzadeh et al.,1995). However, this was negated by Blauvet et al. in 1996 who proved that IL-15 expression is down regulated by UVB in cultured keratinocytes in a dose and time dependent manner (Blauvet et al., 1996).

ELIGIBILITY:
Inclusion criteria:

* Age: ≥ 18 years.
* Both genders.
* Type of Vitiligo: non segmental vitiligo (NSV).
* Active disease for less than 6 months (VIDA ≥ +2).
* No systemic or topical treatment for vitiligo for at least one month.

Exclusion criteria:

* Patients less than 18 years.
* VIDA ≤ +1.
* Contraindications to phototherapy (precancerous conditions like
* Xeroderma pigmentosum , photosensitivity, history of arsenic intake,
* ionizing radiation, extensive previous exposure to PUVA, patients
* with a history of melanoma, atypical nevi, non-melanoma skin
* cancers and patients taking immunosuppressive medications ( Menter et al., 2010 and Mehta & Lim, 2016).
* Pregnancy and lactation .
* Patients who received systemic or topical treatment for the past
* month.
* patients having any autoimmune diseases .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Effect of NB-UVB on tissue level of IL 15 and IL15Rα in active vitiligo | 4 month
  Change of tissue level of Il-15 and IL-15Rα after 48 session of NB-UVB

SECONDARY OUTCOMES:
Effect of activity of vitiligo on tissue level of Il-15 and IL-15Rα | 4 months
  Correlation between tissue level of Il-15 and IL-15Rα before and after NB-UVB with activity score (vitiligo digns of activity score from 0 to 15)
Effect of extent of vitiligo on tissue level of Il-15 and IL-15Rα | 4 month
  Correlation between tissue level of Il-15 and IL-15Rα before and after NB-UVB with extent score (Vitiligo extent plus score )

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan Emad, Principal Investigator — Faculty of medicine kasr Elainy
Locations (1):
- Nourhan Emad, Cairo, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: Yes
I will share the deidentified data sheet of the results of the trial
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 month and ending 12 month after article publication
Access Criteria: Researchers who provide a methodologically sound proposal will be allowed to access the data to achieve aims in the approved proposal Proposal should be directed to nourhanemad693@gmail.com to gain access